CLINICAL TRIAL: NCT02447432
Title: Study to Compare Immunogenicity of GSK Biologicals' 10Pn-PD-DiT 4-dose Presentation to the Licensed Synflorix™ (10Pn-PD-DiT) Vaccine When Co-administered With DTPw-combination Vaccine in Healthy Infants
Brief Title: A Study to Compare the Immunogenicity of GSK Biologicals' 10Pn-PD-DiT 4-dose Presentation to the Licensed 1-dose Synflorix™ (10Pn-PD-DiT) Vaccine When Co-administered With DTPw-combination Vaccine in Healthy Infants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 200799
Record Dates: First submitted 2015-05-07; First posted 2015-05-18 (Estimated); Results first posted 2017-03-16 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-06

CONDITIONS: Infections, Streptococcal
Keywords: Invasive disease by Streptococcus pneumoniae (S. pneumoniae) (including sepsis, meningitis, pneumonia, bacteraemia and acute otitis media); Infants; Multidose; Haemophilus influenzae; Streptococcus pneumoniae; Preservative; Safety; Pneumonia; Immunogenicity; Pneumococcal conjugate vaccine; Acute otitis media caused by non-typeable Haemophilus influenzae (NTHi).; Respiratory tract infections
MeSH Terms: conditions — Streptococcal Infections; Meningitis; Pneumonia; Toxemia; Otitis Media; Haemophilus Infections; Respiratory Tract Infections | interventions — Vaccines; PHiD-CV vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 10Pn_4d Group (Experimental): Subjects received 10Pn-PD-DIT, in its investigational 4-dose presentation (4 doses in total with each single dose injected at Study Months 0, 1, 3 and 8), co administered with DTPw-HBV/Hib vaccine (3 doses injected at Study Months 0, 1 and 2).
  Interventions: Biological: Pneumococcal vaccine GSK1024850A (10Pn-PD-DiT) vaccine (4-dose presentation); Biological: DTPw-HBV/Hib
- 10Pn Group (Active Comparator): Subjects received 10Pn-PD-DIT, in its licensed 1-dose presentation (4 doses in total with each single dose injected at Study Months 0, 1, 3 and 8), co administered with DTPw-HBV/Hib vaccine (3 doses injected at Study Months 0, 1 and 2).
  Interventions: Biological: Pneumococcal vaccine GSK1024850A (10Pn-PD-DiT) vaccine (1-dose presentation); Biological: DTPw-HBV/Hib

INTERVENTIONS:
Biological: Pneumococcal vaccine GSK1024850A (10Pn-PD-DiT) vaccine (4-dose presentation) — 4 doses by intramuscular injection in the right left anterolateral thigh
  Other Names: 10Pn; 10PN-PD-DiT; GSK Biologicals' 10-valent pneumococcal polysaccharide and non-typeable Haemophilus influenzae protein D conjugate GSK1024850A (10Pn-PD-DiT)
  Arms: 10Pn_4d Group
Biological: Pneumococcal vaccine GSK1024850A (10Pn-PD-DiT) vaccine (1-dose presentation) — 4 doses by intramuscular injection in the right anterolateral thigh
  Other Names: Synflorix™; GSK Biologicals' 10-valent pneumococcal polysaccharide and non-typeable Haemophilus influenzae protein D conjugate GSK1024850A (10Pn-PD-DiT) vaccine
  Arms: 10Pn Group
Biological: DTPw-HBV/Hib — 3 doses by intramuscular injection in the left anterolateral thigh
  Other Names: GSK Biologicals' diphtheria-tetanus-whole cell pertussis-hepatitis B and Haemophilus influenzae type b vaccine

SUMMARY:
The primary aim of the study is to demonstrate that an investigational 4-dose presentation of the 10Pn-PD-DiT vaccine with preservative is non-inferior to the licensed presentation of Synflorix (preservative-free) in terms of immune responses to the 10 vaccine pneumococcal serotypes (primary objective) and to the vaccine-related pneumococcal serotype 19A (first secondary objective), after administration of a 3-dose primary vaccination course at 6, 10 and 18 weeks of age co-administered with the first 2 doses of DTPw-HBV/Hib vaccine given at 6, 10 and 14 weeks of age (according to the Expanded Program on Immunization (EPI) schedule).

In addition, the study will also assess the safety, reactogenicity, immunogenicity and antibody persistence (approximately 7 months following primary vaccination) of the 4-dose presentation of the 10Pn-PD-DiT vaccine given as primary vaccination schedule at 6, 10 and 18 weeks of age followed by a booster dose at 38 weeks.

This study also aims at assessing the safety, reactogenicity and immunogenicity of the 4-dose presentation of the 10Pn-PD-DiT vaccine when given as a booster dose at approximately 9 months of age.

ELIGIBILITY:
Inclusion Criteria:

* Subjects for whom, in the opinion of the investigator, the parent(s)/Legally Acceptable Representative(s) [LAR(s)] can and will comply with the requirements of the protocol (e.g., return for vaccination and follow-up visits).
* A male or female between, and including 6-10 weeks (42-76 days) of age at the time of the first vaccination.
* Written or oral, signed or thumb-printed informed consent obtained from the parent(s)/LAR(s) of the subject. For all subjects, the consent form should be countersigned by a witness.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Born full-term (i.e., after a gestation period from 37 to 42 weeks).

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs since birth. Inhaled and topical steroids are allowed.
* Planned administration of long-acting immune-modifying drugs at any time during the study period (e.g., infliximab).
* Administration or planned administration of a vaccine not foreseen by the study protocol administered during the period starting from 30 days before each dose of study vaccines and ending 30 days after with the following exceptions:
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product
* Previous vaccination against diphtheria, tetanus, pertussis, H. influenzae type b and/or S. pneumoniae.
* History of, or intercurrent diphtheria, tetanus, pertussis, hepatitis B, and H. influenzae type b disease.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* Family history of congenital or hereditary immunodeficiency.
* Major congenital defects or serious chronic illness.
* History of any neurological disorders or seizures.
* Acute disease and/or fever at the time of enrolment.
* Fever is defined as temperature ≥ 37.5°C for oral, axillary or tympanic route, or ≥ 38.0°C on rectal route. The preferred route for recording temperature in this study will be axillary.
* Subjects with a minor illness without fever may, be enrolled at the discretion of the investigator.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period (Hepatitis B immunoglobulins at birth are allowed).
* Any medical condition which might interfere with the assessment of the study objectives in the opinion of the investigator.

Ages: 42 Days to 76 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 320 (Actual)
Dates: Start 2015-06-11; Primary Completion 2016-01-23 (Actual); Study Completion 2016-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Zaman K, Zaman SF, Zaman F, Aziz A, Faisal SB, Traskine M, Habib MA, Ruiz-Guinazu J, Borys D. Immunologic non-inferiority and safety of the investigational pneumococcal non-typeable Haemophilus influenzae protein D-conjugate vaccine (PHiD-CV) 4-dose vial presentation compared to the licensed PHiD-CV 1-dose vial presentation in infants: A phase III randomized study. Vaccine. 2018 Jan 29;36(5):698-706. doi: 10.1016/j.vaccine.2017.12.034. Epub 2017 Dec 23. PMID 29277353
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two epochs were defined in the study. The duration of the study was for Epoch 001: Primary starting at Month 0 and ending at Month 4 and for Epoch 002: Booster starting at Month 8 and ending at Month 9. 5 subjects did not participate to the Epoch 002 (none due to an serious adverse event)
Groups:
- 10Pn_4d Group: Healthy male or female subjects between, and including 6 to 10 weeks (42-76 days) of age at the time of first vaccination, received 3 doses of the investigational 4-dose presentation 10Pn-PD-DiT vaccine given approximatively at 6, 10 and 18 weeks of age (primary vaccination - Epoch 001) and 3 doses of DTPw-HBV/Hib vaccine given approximatively at 6, 10 and 14 weeks of age (according to the EPI schedule). They also received a booster dose of the 4-dose presentation 10Pn-PD-DiT vaccine at approximatively 9 months of age (Epoch-002). All vaccines were administered by intramuscular injection in the antero-lateral thigh (10Pn-PD-DiT vaccine: right thigh; DTPw-HBV/Hib vaccine: left thigh).
- Synflorix Group: Healthy male or female subjects between, and including 6 to 10 weeks (42-76 days) of age at the time of first vaccination, received 3 doses of the licensed 1-dose presentation 10Pn-PD-DiT (Synflorix™) vaccine given approximatively at 6, 10 and 18 weeks of age (primary vaccination - Epoch 001) and 3 doses of DTPw-HBV/Hib vaccine given approximatively at 6, 10 and 14 weeks of age (according to the EPI schedule). They also received a booster dose of the 1-dose presentation 10Pn-PD-DiT vaccine at approximatively 9 months of age (Epoch-002). All vaccines were administered by intramuscular injection in the antero-lateral thigh (10Pn-PD-DiT vaccine: right thigh; DTPw-HBV/Hib vaccine: left thigh).
Period: Epoch 001
Arm/Group | 10Pn_4d Group | Synflorix Group
Started | 160 | 160
Completed | 155 | 147
Not Completed | 5 | 13
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Migrated/moved from study area | 3 | 5
Not completed — Lost to Follow-up | 1 | 3
Period: Epoch 002
Arm/Group | 10Pn_4d Group | Synflorix Group
Started | 152 | 145
Completed | 152 | 145
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 10Pn_4d Group: Healthy male or female subjects between, and including 6 to 10 weeks (42-76 days) of age at the time of first vaccination, received 3 doses of the investigational 4-dose presentation 10Pn-PD-DiT vaccine given approximatively at 6, 10 and 18 weeks of age (primary vaccination - Epoch 001) and 3 doses of DTPw-HBV/Hib vaccine given approximatively at 6, 10 and 14 weeks of age (according to the EPI schedule). They also received a booster dose of the 4-dose presentation 10Pn-PD-DiT vaccine at approximatively 9 months of age (Epoch 002). All vaccines were administered by intramuscular injection in the antero-lateral thigh (10Pn-PD-DiT vaccine : right thigh; DTPw-HBV/Hibvaccine : left thigh).
- Synflorix Group: Healthy male or female subjects between, and including 6 to 10 weeks (42-76 days) of age at the time of first vaccination, received 3 doses of the licensed 1-dose presentation 10Pn-PD-DiT (Synflorix™) vaccine given approximatively at 6, 10 and 18 weeks of age (primary vaccination - Epoch 001) and 3 doses of DTPw-HBV/Hib vaccine given approximatively at 6, 10 and 14 weeks of age (according to the EPI schedule). They also received a booster dose of Synflorix™ vaccine at approximatively 9 months of age (Epoch 002). All vaccines were administered by intramuscular injection in the antero-lateral thigh (10Pn-PD-DiT vaccine : right thigh; DTPw-HBV/Hibvaccine : left thigh).
- Total: Total of all reporting groups
Arm/Group | 10Pn_4d Group | Synflorix Group | Total
Number analyzed (Participants) | 160 | 160 | 320
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 6.9 (1.3) | 6.8 (1.2) | 6.8 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 73 | 153
  Male | 80 | 87 | 167
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian-South East Asian heritage | 160 | 160 | 320

OUTCOME MEASURES:

1. Primary Outcome: Antibody Concentrations Against Pneumococcal Serotypes (Epoch 001)
Description: Antibodies assessed for this outcome measure were those against the vaccine/cross-reactive pneumococcal serotypes 1, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F (ANTI-1, -4, -5, -6A, -6B, -7F, -9V, -14, -18C, -19A, -19F and -23F). Antibody concentrations were measured by 22F-inhibition enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL). The cut-off of the assay was an antibody concentration higher than or equal to (≥) 0.05 µg/mL. Primary outcome results correspond to antibody concentrations for the 10 vaccine serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F.
Time Frame: At study Month 4, e. g. at one month post-Dose 3 of pneumococcal vaccine
Population: The analysis was performed on the According To Protocol cohort for immunogenicity of Epoch 001 which included all evaluable subjects (i.e., those meeting eligibility criteria, complied with procedures and intervals defined in protocol, with no elimination criteria) for whom data concerning primary immunogenicity outcomes measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 10Pn_4d Group | Synflorix Group
Number analyzed (Participants) | 154 | 146
µg/mL
  ANTI-1 | 2.78 [2.43 to 3.18] | 3.03 [2.60 to 3.54]
  ANTI-4 | 4.23 [3.69 to 4.84] | 3.87 [3.33 to 4.51]
  ANTI-5 | 5.12 [4.46 to 5.88] | 5.30 [4.59 to 6.12]
  ANTI-6B | 1.23 [0.95 to 1.57] | 1.37 [1.05 to 1.79]
  ANTI-7F | 5.52 [4.90 to 6.22] | 5.79 [5.06 to 6.62]
  ANTI-9V | 4.60 [3.98 to 5.32] | 4.07 [3.34 to 4.95]
  ANTI-14 | 4.97 [4.05 to 6.10] | 4.84 [3.91 to 5.99]
  ANTI-18C | 19.58 [16.65 to 23.03] | 21.18 [17.90 to 25.06]
  ANTI-19F | 13.24 [11.17 to 15.68] | 13.11 [11.16 to 15.41]
  ANTI-23F | 1.59 [1.25 to 2.01] | 2.04 [1.61 to 2.58]
  ANTI-6A | 0.31 [0.25 to 0.38] | 0.29 [0.23 to 0.36]
  ANTI-19A | 0.76 [0.60 to 0.96] | 0.68 [0.54 to 0.86]
Statistical Analysis 1: Comparison: 10Pn_4d Group vs Synflorix Group; (Synflorix/10Pn_4d) antibody GMCs ratio for ANTI-1 serotype: to demonstrate non-inferiority of 10Pn-PD-DiT vaccine (4-dose presentation) as compared to 10Pn-PD-DiT vaccine (1-dose presentation) in terms of immune response, 1 month after dose 3. Criterion: the upper limit (UL) of the 2-sided 95% confidence interval (CI) of the geometric mean antibody concentration (GMC) ratios (Synflorix/10Pn_4d) should be below a limit of 2-fold for each of the 10 serotypes; Test type: Non-Inferiority — GMCs ratio and its 95 % CI were obtained using an ANOVA model on the logarithm-10 transformed concentrations-pooled variance; GMCs ratio = 1.09, 95% CI 2-sided [0.89 to 1.33]
Statistical Analysis 2: Comparison: 10Pn_4d Group vs Synflorix Group; (Synflorix/10Pn_4d) antibody GMCs ratio for ANTI-4 serotype: to demonstrate non-inferiority of 10Pn-PD-DiT vaccine (4-dose presentation) as compared to 10Pn-PD-DiT vaccine (1-dose presentation) in terms of immune response, 1 month after dose 3. Criterion: the upper limit (UL) of the 2-sided 95% confidence interval (CI) of the geometric mean antibody concentration (GMC) ratios (Synflorix/10Pn_4d) should be below a limit of 2-fold for each of the 10 serotypes; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; GMCs ratio = 0.92, 95% CI 2-sided [0.75 to 1.12]
Statistical Analysis 3: Comparison: 10Pn_4d Group vs Synflorix Group; (Synflorix/10Pn_4d) antibody GMCs ratio for ANTI-5 serotype: to demonstrate non-inferiority of 10Pn-PD-DiT vaccine (4-dose presentation) as compared to 10Pn-PD-DiT vaccine (1-dose presentation) in terms of immune response, 1 month after dose 3. Criterion: the upper limit (UL) of the 2-sided 95% confidence interval (CI) of the geometric mean antibody concentration (GMC) ratios (Synflorix/10Pn_4d) should be below a limit of 2-fold for each of the 10 serotypes; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; GMCs ratio = 1.03, 95% CI 2-sided [0.85 to 1.26]
Statistical Analysis 4: Comparison: 10Pn_4d Group vs Synflorix Group; (Synflorix/10Pn_4d) antibody GMCs ratio for ANTI-6B serotype: to demonstrate non-inferiority of 10Pn-PD-DiT vaccine (4-dose presentation) as compared to 10Pn-PD-DiT vaccine (1-dose presentation) in terms of immune response, 1 month after dose 3. Criterion: the upper limit (UL) of the 2-sided 95% confidence interval (CI) of the geometric mean antibody concentration (GMC) ratios (Synflorix/10Pn_4d) should be below a limit of 2-fold for each of the 10 serotypes; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; GMCs ratio = 1.12, 95% CI 2-sided [0.78 to 1.61]
Statistical Analysis 5: Comparison: 10Pn_4d Group vs Synflorix Group; (Synflorix/10Pn_4d) antibody GMCs ratio for ANTI-7F serotype: to demonstrate non-inferiority of 10Pn-PD-DiT vaccine (4-dose presentation) as compared to 10Pn-PD-DiT vaccine (1-dose presentation) in terms of immune response, 1 month after dose 3. Criterion: the upper limit (UL) of the 2-sided 95% confidence interval (CI) of the geometric mean antibody concentration (GMC) ratios (Synflorix/10Pn_4d) should be below a limit of 2-fold for each of the 10 serotypes; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; GMCs ratio = 1.05, 95% CI 2-sided [0.88 to 1.25]
Statistical Analysis 6: Comparison: 10Pn_4d Group vs Synflorix Group; (Synflorix/10Pn_4d) antibody GMCs ratio for ANTI-9V serotype: to demonstrate non-inferiority of 10Pn-PD-DiT vaccine (4-dose presentation) as compared to 10Pn-PD-DiT vaccine (1-dose presentation) in terms of immune response, 1 month after dose 3. Criterion: the upper limit (UL) of the 2-sided 95% confidence interval (CI) of the geometric mean antibody concentration (GMC) ratios (Synflorix/10Pn_4d) should be below a limit of 2-fold for each of the 10 serotypes; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; GMCs ratio = 0.88, 95% CI 2-sided [0.69 to 1.13]
Statistical Analysis 7: Comparison: 10Pn_4d Group vs Synflorix Group; (Synflorix/10Pn_4d) antibody GMCs ratio for ANTI-14 serotype: to demonstrate non-inferiority of 10Pn-PD-DiT vaccine (4-dose presentation) as compared to 10Pn-PD-DiT vaccine (1-dose presentation) in terms of immune response, 1 month after dose 3. Criterion: the upper limit (UL) of the 2-sided 95% confidence interval (CI) of the geometric mean antibody concentration (GMC) ratios (Synflorix/10Pn_4d) should be below a limit of 2-fold for each of the 10 serotypes; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; GMCs ratio = 0.98, 95% CI 2-sided [0.73 to 1.31]
Statistical Analysis 8: Comparison: 10Pn_4d Group vs Synflorix Group; (Synflorix/10Pn_4d) antibody GMCs ratio for ANTI-18C serotype: to demonstrate non-inferiority of 10Pn-PD-DiT vaccine (4-dose presentation) as compared to 10Pn-PD-DiT vaccine (1-dose presentation) in terms of immune response, 1 month after dose 3. Criterion: the upper limit (UL) of the 2-sided 95% confidence interval (CI) of the geometric mean antibody concentration (GMC) ratios (Synflorix/10Pn_4d) should be below a limit of 2-fold for each of the 10 serotypes; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; GMCs ratio = 1.08, 95% CI 2-sided [0.86 to 1.37]
Statistical Analysis 9: Comparison: 10Pn_4d Group vs Synflorix Group; (Synflorix/10Pn_4d) antibody GMCs ratio for ANTI-19F serotype: to demonstrate non-inferiority of 10Pn-PD-DiT vaccine (4-dose presentation) as compared to 10Pn-PD-DiT vaccine (1-dose presentation) in terms of immune response, 1 month after dose 3. Criterion: the upper limit (UL) of the 2-sided 95% confidence interval (CI) of the geometric mean antibody concentration (GMC) ratios (Synflorix/10Pn_4d) should be below a limit of 2-fold for each of the 10 serotypes; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; GMCs ratio = 0.99, 95% CI 2-sided [0.78 to 1.25]
Statistical Analysis 10: Comparison: 10Pn_4d Group vs Synflorix Group; (Synflorix/10Pn_4d) antibody GMCs ratio for ANTI-23F serotype: to demonstrate non-inferiority of 10Pn-PD-DiT vaccine (4-dose presentation) as compared to 10Pn-PD-DiT vaccine (1-dose presentation) in terms of immune response, 1 month after dose 3. Criterion: the upper limit (UL) of the 2-sided 95% confidence interval (CI) of the geometric mean antibody concentration (GMC) ratios (Synflorix/10Pn_4d) should be below a limit of 2-fold for each of the 10 serotypes; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; GMCs ratio = 1.28, 95% CI 2-sided [0.92 to 1.80]

2. Secondary Outcome: Antibody Concentrations Against Pneumococcal Serotypes (Epoch 002)
Description: Antibodies assessed for this outcome measure were those against the vaccine/cross-reactive pneumococcal serotypes 1, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F (ANTI-1, -4, -5, -6A, -6B, -7F, -9V, -14, -18C, -19A, -19F and -23F). Antibody concentrations were measured by 22F-inhibition enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in micrograms per milliliter (µg/mL). The cut-off of the assay was an antibody concentration higher than or equal to (≥) 0.05 µg/mL.
Time Frame: At Month 8 and Month 9, e.g.: prior to and at one month post booster vaccination with pneumococcal vaccine
Population: The analysis was performed on the According To Protocol cohort for immunogenicity of Epoch 002 which included all evaluable subjects (i.e., those meeting eligibility criteria, complied with procedures and intervals defined in protocol, with no elimination criteria) for whom data concerning booster immunogenicity outcomes measures were available.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | 10Pn_4d Group | Synflorix Group
Number analyzed (Participants) | 151 | 144
µg/mL
  ANTI-1 Month 8 | 0.93 [0.79 to 1.1] | 0.99 [0.81 to 1.19]
  ANTI-1 Month 9 | 6.37 [5.48 to 7.41] | 7.5 [6.28 to 8.97]
  ANTI-4 Month 8 | 1.9 [1.65 to 2.19] | 1.71 [1.45 to 2.01]
  ANTI-4 Month 9: number analyzed (Participants) | 151 | 143
  ANTI-4 Month 9 | 9.68 [8.47 to 11.06] | 9.41 [8.16 to 10.86]
  ANTI-5 Month 8 | 1.75 [1.5 to 2.05] | 1.75 [1.48 to 2.08]
  ANTI-5 Month 9 | 11.53 [10.14 to 13.12] | 12.24 [10.65 to 14.05]
  ANTI-6B Month 8 | 1.14 [0.93 to 1.4] | 1.06 [0.84 to 1.32]
  ANTI-6B Month 9 | 3.76 [3.01 to 4.69] | 4.11 [3.21 to 5.25]
  ANTI-7F Month 8 | 2.86 [2.5 to 3.27] | 2.75 [2.4 to 3.16]
  ANTI-7F Month 9 | 12.84 [11.38 to 14.48] | 13.71 [12.01 to 15.65]
  ANTI-9V Month 8 | 2.32 [1.96 to 2.75] | 2.25 [1.83 to 2.76]
  ANTI-9V Month 9 | 12.07 [10.42 to 13.98] | 12.43 [10.22 to 15.13]
  ANTI-14 Month 8 | 2.98 [2.39 to 3.72] | 2.4 [1.9 to 3.04]
  ANTI-14 Month 9: number analyzed (Participants) | 151 | 143
  ANTI-14 Month 9 | 9.84 [8.02 to 12.08] | 9.72 [7.92 to 11.93]
  ANTI-18C Month 8 | 8.37 [7.14 to 9.82] | 9.23 [7.82 to 10.9]
  ANTI-18C Month 9 | 41.64 [36.87 to 47.02] | 47.06 [41.88 to 52.88]
  ANTI-19F Month 8 | 6.36 [5.36 to 7.55] | 6.45 [5.5 to 7.57]
  ANTI-19F Month 9 | 23.43 [19.48 to 28.19] | 24.96 [21.07 to 29.57]
  ANTI-23F Month 8 | 1.09 [0.89 to 1.33] | 1.21 [0.96 to 1.53]
  ANTI-23F Month 9 | 6.69 [5.66 to 7.9] | 6.69 [5.33 to 8.41]
  ANTI-6A Month 8 | 0.31 [0.24 to 0.39] | 0.3 [0.24 to 0.38]
  ANTI-6A Month 9 | 0.97 [0.74 to 1.26] | 1.11 [0.83 to 1.49]
  ANTI-19A Month 8 | 0.7 [0.55 to 0.89] | 0.69 [0.54 to 0.88]
  ANTI-19A Month 9 | 3.03 [2.26 to 4.05] | 3.63 [2.73 to 4.82]

3. Secondary Outcome: Titers for Opsonophagocytic Activity Against Pneumococcal Serotypes (Epoch 001)
Description: Titers for opsonophagocytic activity assessed for this outcome measure were those for opsonophagocytic activity against the vaccine/cross-reactive pneumococcal serotypes 1, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F (OPA-1, -4, -5, -6A, -6B, -7F, -9V, -14, -18C, 19 A ,-19F and -23F). The cut-off of the assay was a titer for opsonophagocytic activity higher than or equal to (≥) 8.
Time Frame: At study Month 4, e. g. at one month post-Dose 3 of pneumococcal vaccine
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 10Pn_4d Group | Synflorix Group
Number analyzed (Participants) | 75 | 74
Titers
  OPA-1: number analyzed (Participants) | 74 | 74
  OPA-1 | 48.3 [34.9 to 67.0] | 52.8 [36.0 to 77.5]
  OPA-4 | 823.1 [670.9 to 1009.8] | 836.8 [644.5 to 1086.6]
  OPA-5: number analyzed (Participants) | 73 | 74
  OPA-5 | 179.0 [140.7 to 227.8] | 211.0 [162.9 to 273.2]
  OPA-6B: number analyzed (Participants) | 73 | 73
  OPA-6B | 560.6 [336.9 to 932.8] | 759.6 [470.2 to 1227.3]
  OPA-7F: number analyzed (Participants) | 74 | 73
  OPA-7F | 2044.0 [1669.3 to 2502.9] | 2076.8 [1627.0 to 2650.9]
  OPA-9V | 613.3 [444.9 to 845.4] | 821.1 [602.5 to 1119.2]
  OPA-14: number analyzed (Participants) | 73 | 74
  OPA-14 | 1563.9 [1105.1 to 2213.2] | 1655.8 [1141.1 to 2402.7]
  OPA-18C | 3965.4 [3288.6 to 4781.5] | 3809.7 [3067.0 to 4732.3]
  OPA-19F | 2151.3 [1573.5 to 2941.4] | 2879.2 [2348.4 to 3529.9]
  OPA-23F | 524.8 [338.5 to 813.9] | 730.2 [495.6 to 1075.7]
  OPA-6A: number analyzed (Participants) | 66 | 69
  OPA-6A | 50.3 [26.9 to 94.0] | 68.5 [36.8 to 127.7]
  OPA-19A: number analyzed (Participants) | 72 | 71
  OPA-19A | 98.6 [60.9 to 159.6] | 117.1 [71.9 to 190.6]

4. Secondary Outcome: Titers for Opsonophagocytic Activity Against Pneumococcal Serotypes (Epoch 002)
Description: Titers for opsonophagocytic activity assessed for this outcome measure were those for opsonophagocytic activity against the vaccine/cross-reactive pneumococcal serotypes 1, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F (OPA-1, -4, -5, -6A, -6B, -7F, -9V, -14, -18C, -19A, -19F and -23F). The cut-off of the assay was a titer for opsonophagocytic activity higher than or equal to (≥) 8.
Time Frame: At study Month 8 and Month 9, e.g.: prior to and at one month post booster vaccination with pneumococcal vaccine
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | 10Pn_4d Group | Synflorix Group
Number analyzed (Participants) | 76 | 73
Titers
  OPA-1 Month 8: number analyzed (Participants) | 72 | 70
  OPA-1 Month 8 | 11.5 [8.2 to 16.1] | 12.8 [9.1 to 17.9]
  OPA-1 Month 9: number analyzed (Participants) | 73 | 71
  OPA-1 Month 9 | 227.7 [170.6 to 303.9] | 326.7 [238.7 to 447]
  OPA-4 Month 8: number analyzed (Participants) | 72 | 70
  OPA-4 Month 8 | 248.1 [178.6 to 344.7] | 280.5 [193.4 to 406.6]
  OPA-4 Month 9 | 2025.4 [1641.6 to 2498.8] | 2888.7 [2221.6 to 3756.1]
  OPA-5 Month 8: number analyzed (Participants) | 73 | 71
  OPA-5 Month 8 | 51.3 [37 to 71.3] | 62.7 [44.4 to 88.7]
  OPA-5 Month 9 | 550.6 [437.8 to 692.4] | 801.2 [633.2 to 1013.6]
  OPA-6B Month 8: number analyzed (Participants) | 73 | 70
  OPA-6B Month 8 | 290.3 [177.1 to 475.7] | 286.8 [183.5 to 448]
  OPA-6B Month 9: number analyzed (Participants) | 74 | 72
  OPA-6B Month 9 | 851.3 [533.4 to 1358.6] | 1352 [913.9 to 1999.9]
  OPA-7F Month 8: number analyzed (Participants) | 74 | 73
  OPA-7F Month 8 | 1112.8 [864.8 to 1431.8] | 1181.7 [933.4 to 1495.9]
  OPA-7F Month 9 | 4574.7 [3756.1 to 5571.6] | 5635.8 [4561.7 to 6962.9]
  OPA-9V Month 8: number analyzed (Participants) | 69 | 72
  OPA-9V Month 8 | 415.8 [280.6 to 616.3] | 570.6 [408.4 to 797.3]
  OPA-9V Month 9 | 2308.4 [1903.3 to 2799.7] | 3181.9 [2376.9 to 4259.6]
  OPA-14 Month 8: number analyzed (Participants) | 73 | 72
  OPA-14 Month 8 | 660.1 [432.4 to 1007.6] | 745 [513.9 to 1080]
  OPA-14 Month 9 | 3345.6 [2585 to 4330.1] | 3649.1 [2808.6 to 4741.2]
  OPA-18C Month 8: number analyzed (Participants) | 74 | 73
  OPA-18C Month 8 | 1505.4 [1196.4 to 1894.1] | 1735.2 [1373.8 to 2191.7]
  OPA-18C Month 9 | 7316.1 [6137.6 to 8720.8] | 7181.6 [6003.6 to 8590.7]
  OPA-19F Month 8: number analyzed (Participants) | 74 | 72
  OPA-19F Month 8 | 770.1 [536.6 to 1105.3] | 1254.3 [990.8 to 1587.9]
  OPA-19F Month 9 | 3197.3 [2271.1 to 4501.2] | 4757.7 [3772.3 to 6000.4]
  OPA-23F Month 8: number analyzed (Participants) | 70 | 69
  OPA-23F Month 8 | 267.7 [168.7 to 424.9] | 252.7 [154.8 to 412.4]
  OPA-23F Month 9 | 1250.8 [931.3 to 1679.8] | 1465.6 [1002.9 to 2141.7]
  OPA-6A Month 8: number analyzed (Participants) | 72 | 68
  OPA-6A Month 8 | 52.4 [27.4 to 100.1] | 45.5 [24 to 86.5]
  OPA-6A Month 9: number analyzed (Participants) | 71 | 68
  OPA-6A Month 9 | 192 [102.9 to 358.4] | 284.4 [158.4 to 510.6]
  OPA-19A Month 8: number analyzed (Participants) | 73 | 71
  OPA-19A Month 8 | 42.7 [25.1 to 72.7] | 43.6 [26.6 to 71.3]
  OPA-19A Month 9: number analyzed (Participants) | 76 | 72
  OPA-19A Month 9 | 410.4 [246.7 to 682.8] | 591.7 [356.9 to 980.9]

5. Secondary Outcome: Concentrations of Antibodies Against Protein D (Anti-PD) (Epoch 001)
Description: Anti-PD antibody concentrations were measured by enzyme-linked immunosorbent assay (ELISA), expressed as geometric mean concentrations (GMCs), in ELISA Units per milliliter (EL.U/mL). The cut-off of the assay was an anti-PD antibody concentration higher than or equal to (≥) 153 EL.U/mL.
Time Frame: At study Month 4, e. g. at one month post-Dose 3 of pneumococcal vaccine
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | 10Pn_4d Group | Synflorix Group
Number analyzed (Participants) | 78 | 75
EL.U/mL | 2410.5 [2029.2 to 2863.5] | 2495.4 [2055.7 to 3029.1]

6. Secondary Outcome: Concentrations of Antibodies Against Protein D (Anti-PD) (Epoch 002)
Description: as for outcome 5
Time Frame: At study Month 9, e.g.: at one month post booster vaccination with pneumococcal vaccine
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | 10Pn_4d Group | Synflorix Group
Number analyzed (Participants) | 76 | 73
EL.U/mL | 2672.4 [2285.5 to 3124.8] | 2944 [2486.2 to 3486]

7. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms (Epoch 001)
Description: Assessed local symptoms were pain, redness and swelling. Any = Occurrence of the specified solicited local symptom, regardless of intensity. Grade 3 Pain = Crying when limb was moved/spontaneously painful. Grade 3 Redness/Swelling = Redness/swelling at injection site larger than (>) 30 millimeters (mm). Dose 1 = 10Pn-PD-DIT+DTPw-HBV/Hib at 6 weeks of age. Dose 2 = 10Pn-PD-DIT+DTPw-HBV/Hib at 10 weeks of age.
  Dose 4 = 10Pn-PD-DIT at 18 weeks of age.
Time Frame: Within the 4-day (Days 0-3) post-vaccination period following each primary dose of 10Pn-PD-DiTvaccine
Population: The analysis was performed on the Total vaccinated cohort of Epoch 001 included all subjects who had received at least one dose of primary vaccination, with analysis done solely on subjects for whom post-vaccination results about solicited symptoms were available.
Measure: Count of Participants; unit: Participants
Arm/Group | 10Pn_4d Group | Synflorix Group
Number analyzed (Participants) | 159 | 156
Participants
  Any Pain, post Dose 1 | 82 | 90
  Grade 3 Pain, post Dose 1 | 4 | 5
  Any Redness, post Dose 1 | 24 | 26
  Grade 3 Redness, post Dose 1 | 0 | 0
  Any Swelling, post Dose 1 | 63 | 64
  Grade 3 Swelling, post Dose 1 | 0 | 0
  Any Pain, post Dose 2: number analyzed (Participants) | 158 | 152
  Any Pain, post Dose 2 | 56 | 56
  Grade 3 Pain, post Dose 2: number analyzed (Participants) | 158 | 152
  Grade 3 Pain, post Dose 2 | 1 | 0
  Any Redness, post Dose 2: number analyzed (Participants) | 158 | 152
  Any Redness, post Dose 2 | 22 | 26
  Grade 3 Redness, post Dose 2: number analyzed (Participants) | 158 | 152
  Grade 3 Redness, post Dose 2 | 0 | 0
  Any Swelling, post Dose 2: number analyzed (Participants) | 158 | 152
  Any Swelling, post Dose 2 | 31 | 37
  Grade 3 Swelling, post Dose 2: number analyzed (Participants) | 158 | 152
  Grade 3 Swelling, post Dose 2 | 0 | 0
  Any Pain, post Dose 4: number analyzed (Participants) | 155 | 147
  Any Pain, post Dose 4 | 13 | 15
  Grade 3 Pain, post Dose 4: number analyzed (Participants) | 155 | 147
  Grade 3 Pain, post Dose 4 | 0 | 0
  Any Redness, post Dose 4: number analyzed (Participants) | 155 | 147
  Any Redness, post Dose 4 | 9 | 8
  Grade 3 Redness, post Dose 4: number analyzed (Participants) | 155 | 147
  Grade 3 Redness, post Dose 4 | 0 | 0
  Any Swelling, post Dose 4: number analyzed (Participants) | 155 | 147
  Any Swelling, post Dose 4 | 11 | 9
  Grade 3 Swelling, post Dose 4: number analyzed (Participants) | 155 | 147
  Grade 3 Swelling, post Dose 4 | 0 | 0

8. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms (Epoch 002)
Description: Assessed local symptoms were pain, redness and swelling. Any = Occurrence of the specified solicited local symptom, regardless of intensity. Grade 3 Pain = Crying when limb was moved/spontaneously painful. Grade 3 Redness/Swelling = Redness/swelling at injection site larger than (>) 30 millimeters (mm).
Time Frame: Within the 4-day (Days 0-3) period after booster vaccination
Population: The analysis was performed on the Total vaccinated cohort of Epoch 002 included all subjects who had received the booster vaccination, with analysis done solely on subjects for whom post-vaccination results about solicited or unsolicited symptoms were available.
Measure: Count of Participants; unit: Participants
Arm/Group | 10Pn_4d Group | Synflorix Group
Number analyzed (Participants) | 152 | 145
Participants
  Any Pain | 9 | 2
  Grade 3 Pain | 1 | 0
  Any Redness | 14 | 5
  Grade 3 Redness | 0 | 0
  Any Swelling | 16 | 8
  Grade 3 Swelling | 0 | 0

9. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited General Symptoms and With Solicited General Symptoms With Relationship to Vaccination(Epoch 001)
Description: Assessed solicited general symptoms were Drowsiness, Irritability/Fussiness, Loss of appetite and Fever (axillary route - temperature equal or higher than [≥] 37.5 degrees Celsius [°C]). Any = Occurrence of the specified solicited general symptom, regardless of intensity or relationship to vaccination. Grade 3 Drowsiness = Drowsiness that prevented normal activity. Grade 3 Irritability/Fussiness = Crying that could not be comforted/prevented normal activity. Grade 3 Loss of appetite = Subject did not eat at all. Grade 3 Fever = (axillary) temperature higher than (>) 39.5°C. Related = Occurrence of the specified symptom assessed by the investigator as causally related to vaccination. Dose 1 = 10Pn-PD-DIT+DTPw-HBV/Hib at 6 weeks of age. Dose 2 = 10Pn-PD-DIT+DTPw-HBV/Hib at 10 weeks of age.
  Dose 4 = 10Pn-PD-DIT at 18 weeks of age.
Time Frame: Within the 4-day (Days 0-3) post-vaccination period following each primary dose of 10Pn-PD-DiTvaccine
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | 10Pn_4d Group | Synflorix Group
Number analyzed (Participants) | 159 | 156
Participants
  Any Drowsiness, post Dose 1 | 26 | 31
  Grade 3 Drowsiness, post Dose 1 | 1 | 5
  Related Drowsiness, post Dose 1 | 26 | 29
  Any Irritability/Fussiness, post Dose 1 | 61 | 62
  Grade 3 Irritability/Fussiness, post Dose 1 | 14 | 8
  Related Irritability/Fussiness, post Dose 1 | 61 | 62
  Any Loss Appetite, post Dose 1 | 43 | 46
  Grade 3 Loss Appetite, post Dose 1 | 4 | 3
  Related Loss Appetite, post Dose 1 | 43 | 46
  Any Fever, post Dose 1 | 28 | 30
  Grade 3 Fever, post Dose 1 | 0 | 0
  Related Fever, post Dose 1 | 28 | 30
  Any Drowsiness, post Dose 2: number analyzed (Participants) | 158 | 152
  Any Drowsiness, post Dose 2 | 15 | 23
  Grade 3 Drowsiness, post Dose 2: number analyzed (Participants) | 158 | 152
  Grade 3 Drowsiness, post Dose 2 | 1 | 1
  Related Drowsiness, post Dose 2: number analyzed (Participants) | 158 | 152
  Related Drowsiness, post Dose 2 | 15 | 23
  Any Irritability/Fussiness, post Dose 2: number analyzed (Participants) | 158 | 152
  Any Irritability/Fussiness, post Dose 2 | 39 | 47
  Grade 3 Irritability/Fussiness, post D2: number analyzed (Participants) | 158 | 152
  Grade 3 Irritability/Fussiness, post D2 | 4 | 5
  Related Irritability/Fussiness, post Dose 2: number analyzed (Participants) | 158 | 152
  Related Irritability/Fussiness, post Dose 2 | 39 | 47
  Any Loss Appetite, post Dose 2: number analyzed (Participants) | 158 | 152
  Any Loss Appetite, post Dose 2 | 24 | 20
  Grade 3 Loss Appetite, post Dose 2: number analyzed (Participants) | 158 | 152
  Grade 3 Loss Appetite, post Dose 2 | 3 | 2
  Related Loss Appetite, post Dose 2: number analyzed (Participants) | 158 | 152
  Related Loss Appetite, post Dose 2 | 23 | 20
  Any Fever, post Dose 2: number analyzed (Participants) | 158 | 152
  Any Fever, post Dose 2 | 23 | 18
  Grade 3 Fever, post Dose 2: number analyzed (Participants) | 158 | 152
  Grade 3 Fever, post Dose 2 | 0 | 0
  Related Fever, post Dose 2: number analyzed (Participants) | 158 | 152
  Related Fever, post Dose 2 | 22 | 18
  Any Drowsiness, post Dose 4: number analyzed (Participants) | 155 | 147
  Any Drowsiness, post Dose 4 | 6 | 8
  Grade 3 Drowsiness, post Dose 4: number analyzed (Participants) | 155 | 147
  Grade 3 Drowsiness, post Dose 4 | 0 | 1
  Related Drowsiness, post Dose 4: number analyzed (Participants) | 155 | 147
  Related Drowsiness, post Dose 4 | 6 | 8
  Any Irritability/Fussiness, post Dose 4: number analyzed (Participants) | 155 | 147
  Any Irritability/Fussiness, post Dose 4 | 10 | 12
  Grade 3 Irritability/Fussiness, post Dose 4: number analyzed (Participants) | 155 | 147
  Grade 3 Irritability/Fussiness, post Dose 4 | 0 | 1
  Related Irritability/Fussiness, post Dose 4: number analyzed (Participants) | 155 | 147
  Related Irritability/Fussiness, post Dose 4 | 10 | 12
  Any Loss Appetite, post Dose 4: number analyzed (Participants) | 155 | 147
  Any Loss Appetite, post Dose 4 | 5 | 5
  Grade 3 Loss Appetite, post Dose 4: number analyzed (Participants) | 155 | 147
  Grade 3 Loss Appetite, post Dose 4 | 0 | 0
  Related Loss Appetite, post Dose 4: number analyzed (Participants) | 155 | 147
  Related Loss Appetite, post Dose 4 | 5 | 5
  Any Fever, post Dose 4: number analyzed (Participants) | 155 | 147
  Any Fever, post Dose 4 | 2 | 6
  Grade 3 Fever, post Dose 4: number analyzed (Participants) | 155 | 147
  Grade 3 Fever, post Dose 4 | 0 | 0
  Related Fever, post Dose 4: number analyzed (Participants) | 155 | 147
  Related Fever, post Dose 4 | 2 | 6

10. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited General Symptoms and With Solicited General Symptoms With Relationship to Vaccination (Epoch 002)
Description: Assessed solicited general symptoms were Drowsiness, Irritability/Fussiness, Loss of appetite and Fever (axillary route - temperature equal or higher than [≥] 37.5 degrees Celsius [°C]). Any = Occurrence of the specified solicited general symptom, regardless of intensity or relationship to vaccination. Related = Occurrence of the specified symptom assessed by the investigators as causally related to vaccination. Grade 3 Drowsiness = Drowsiness that prevented normal activity. Grade 3 Irritability/Fussiness = Crying that could not be comforted/prevented normal activity. Grade 3 Loss of appetite = Subject did not eat at all. Grade 3 Fever = (Axillary) temperature higher than (>) 39.5°C.
Time Frame: Within the 4-day (Days 0-3) period after booster vaccination
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | 10Pn_4d Group | Synflorix Group
Number analyzed (Participants) | 152 | 145
Participants
  Any Drowsiness | 8 | 4
  Grade 3 Drowsiness | 0 | 0
  Related Drowsiness | 8 | 4
  Any Irritability/Fussiness | 11 | 5
  Grade 3 Irritability/Fusiness | 1 | 0
  Related Irritability/Fussiness | 11 | 5
  Any Loss Appetite | 8 | 4
  Grade 3 Loss Appetite | 0 | 0
  Related Loss Appetite | 8 | 4
  Any Fever | 4 | 3
  Grade 3 Fever | 0 | 0
  Related Fever | 4 | 3

11. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs) (Epoch 001)
Description: An unsolicited AE was defined as any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. For the marketed products administered in the study, this also included failure to produce expected benefits (i.e. lack of efficacy), abuse or misuse of the product. Any = Occurrence of an unsolicited AE, regardless of intensity or relationship to vaccination.
Time Frame: Within the 31-day (Days 0-30) period post primary vaccination, across doses
Population: The analysis was performed on the Total vaccinated cohort of Epoch 001 which included all subjects who had received at least one dose of primary vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 10Pn_4d Group | Synflorix Group
Number analyzed (Participants) | 160 | 160
Participants | 10 | 16

12. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs) (Epoch 002)
Description: as for outcome 11
Time Frame: Within the 31-day (Days 0-30) period post booster vaccination
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | 10Pn_4d Group | Synflorix Group
Number analyzed (Participants) | 152 | 145
Participants | 0 | 0

13. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs) (Epoch 001)
Description: An SAE was defined as any medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity in a subject. AE(s) considered as SAE(s) also included invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that did not result in hospitalization, as per the medical or scientific judgement of the physician. Any = Occurrence of an SAE, regardless of relationship to vaccination.
Time Frame: From Month 0 to Month 4
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | 10Pn_4d Group | Synflorix Group
Number analyzed (Participants) | 160 | 160
Participants | 4 | 9

14. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs) During the Entire Duration of the Study
Description: as for outcome 13
Time Frame: From Day 0 to Month 9
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | 10Pn_4d Group | Synflorix Group
Number analyzed (Participants) | 160 | 160
Participants | 4 | 9

ADVERSE EVENTS:
Time Frame: Solicited symptoms and Unsolicited AEs: during 31 days post vaccination period. SAEs: during the whole study period (from Day 0 to Month 9).
Arm/Group | 10Pn_4d Group | Synflorix Group
All-Cause Mortality (participants affected / at risk) | 1/160 | 1/160
Serious Adverse Events (participants affected / at risk) | 4/160 | 9/160
Other Adverse Events (participants affected / at risk) | 120/160 | 126/160
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10Pn_4d Group (N=160) | Synflorix Group (N=160)
Cerebral palsy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Laryngomalacia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (3)
Bronchiolitis (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 4 (4)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Chemical poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10Pn_4d Group (N=160) | Synflorix Group (N=160)
Pain (General disorders) | 101 (160) | 102 (163)
Pyrexia (General disorders) | 51 (59) | 47 (57)
Swelling (General disorders) | 83 (121) | 81 (118)
Decreased appetite (Metabolism and nutrition disorders) | 58 (80) | 53 (75)
Somnolence (Nervous system disorders) | 38 (55) | 42 (66)
Irritability (Psychiatric disorders) | 77 (121) | 84 (126)
Erythema (Skin and subcutaneous tissue disorders) | 37 (69) | 40 (65)

LIMITATIONS AND CAVEATS:
None reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.